CLINICAL TRIAL: NCT03558815
Title: Psychotropic Medication and Psychotherapeutic Treatment of Adults With Intellectual Disabilities
Acronym: PROMPT-ID
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Matthias Schützwohl, Head of Mental Health Services Research Group, Technische Universität Dresden
Other Study IDs: 040_5121
Record Dates: First submitted 2018-05-15; First posted 2018-06-15 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Intellectual Disability
Keywords: intellectual disability; psychotropic medication; mental health services evaluation
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with mild, moderate, severe or profound ID: Adults with mild, moderate, severe or profound ID in contact with either a sheltered workshop and/ or sheltered living Institution in Saxony.

SUMMARY:
Mental health service provision of adults with intellectual disabilities (ID) is often criticized. There is a lack of empirically studies targeting the psychotropic and psychotherapeutic treatment in this population. The PROMPT-ID study therefore aims to assess the prevalence of psychotropic medication and psychotherapeutic treatment in adults with mild to profound ID and the quality of psychotropic medication. It further aims to identify predictors of psychotropic medication, of barriers into psychotherapeutic treatment and of good clinical psychotropic medication prescription practice. It is a cross-sectional, epidemiological study carried out in Saxony, Germany. Approval of the responsible ethics committee was obtained. The inclusion criteria are mild to profound forms of ID and an age of 18 years or older. A representative sample is realized by a two-stage sampling procedure. Sheltered working and accommodation service providers are stratified by type of service provider and workshop size/type of accommodation. The stratified cluster sampling is realized by a random selection of service providing institutions followed by a random selection of adults with ID. An estimated total number of n = 200 study participants via sheltered workshops and n = 400 via residential accommodations need to be contacted to obtain data of approximately n = 131 study participants recruited through sheltered workshops and n = 232 participants through sheltered living institutions. Based on a psychotropic medication prevalence of 30%, in- depth interviews about psychotropic prescription practice of an estimated number of n = 109 adults with ID are carried out. Data collection is realized in interviews with key carers in the living environment and, if applicable, with the prescribing physician. If the adults with ID are currently medicated with psychotropics, basic information e.g. about kind, agent, dosage and treatment duration are obtained and a newly developed interview targeting the quality of the psychotropic medication treatment is conducted with the carers. In addition to the prevalence and quality of psychotropic and psychotherapeutic health care utilisation, other parameters like psychiatric symptomatology, problem behavior, sociodemografic and institutional factors and parameters of the provision area are assessed using well- established instruments. Findings will fill the lack of representative data that is urgently needed in this often criticized health service area.

ELIGIBILITY:
Inclusion Criteria:

* Mild to profound levels of ID
* Age of 18 years or older

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are adults with mild to profound levels of intellectual disability using sheltered working and/or sheltered accommodation services.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Quality of psychotropic medication (Interview for Assessing the Quality of Psychopharmacological Treatment of Adults with Intellectual Disabilities (IQP-ID; Schützwohl et al., 2017) | 3 months
  If the adults with ID had a psychotropic medication prescription of at least one of the following six substance classes in the past three months: neuroleptics, antidepressants, benzodiazepines, lithium, anxiolytics/sedatives and/or antiepileptics, the Interview for Assessing the Quality of Psychopharmacological Treatment of Adults with Intellectual Disabilities (IQP-ID; Schützwohl et al., 2017) is conducted. This interview assesses the prescription practice of psychotropic medication in adults with ID. It is based on current guidelines of psychotropic medication prescription in adults with ID.The interview comprises 13 quality indicators that are assigned to one of 7 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schützwohl, Prof. Dr., Principal Investigator — Department of Psychiatry and Psychoptherapy
Locations (1):
- Department of psychiatry and Psychotherapy, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koch A, Dobrindt J, Schutzwohl M. Psychotropic medication and psychotherapeutic treatment of adults with intellectual disabilities (PROMPT-ID): a cross-sectional, epidemiological study in Saxony, Germany. BMJ Open. 2018 Dec 19;8(12):e025947. doi: 10.1136/bmjopen-2018-025947. PMID 30573492